CLINICAL TRIAL: NCT05807711
Title: Efficacy of L-methylfolate and Methylcobalamine in Treating Resistant Hypertension Associated with Elevated Serum Homocysteine in Hemodialysis Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107591
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2023-03

CONDITIONS: End Stage Renal Disease; Hypertension, Renal
Keywords: L-methylfolate; methylcobalamine; homocysteine
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension, Renal | interventions — 5-methyltetrahydrofolate; mecobalamin

STUDY DESIGN:
Intervention Model Description: open-label, single-center, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Intervention group (Active Comparator): Adult end stage renal disease patients maintained on hemodialysis three times a week for at least 3 months with resistant hypertension as determined by pre-dialysis BP > 140/90 mm Hg, post-dialysis BP > 130/80 mm Hg despite the use of three or more drugs.
  Patients will be assigned to take one tablet daily containing L-methylfolate and methylcobalamine.
  Patients will be followed over a period of 3 months after which blood pressure measurement and blood sampling would be repeated and compared to baseline values.
  Interventions: Drug: L-Methyl Folate and methylcobalamine
- No Intervention: Control group (No Intervention): Adult end stage renal disease patients maintained on hemodialysis three times a week for at least 3 months with resistant hypertension as determined by pre-dialysis BP > 140/90 mm Hg, post-dialysis BP > 130/80 mm Hg despite the use of three or more drugs.
  Patients will be followed over a period of 3 months after which blood pressure measurement and blood sampling would be repeated and compared to baseline values.

INTERVENTIONS:
Drug: L-Methyl Folate and methylcobalamine — Dietary supplement labeled to contain methylfolate 800 micrograms and methylcobalamine 1000 micrograms
  Arms: Experimental: Intervention group

SUMMARY:
The aim of the study is to evaluate the efficacy of L-methylfolate in combination with methylcobalamine in reducing homocysteine blood levels in hypertensive end-stage renal disease patients on regular hemodialysis and its association with blood pressure control in treatment of resistant hypertension

DETAILED DESCRIPTION:
1. Ethical committee approval has been obtained from Ethics committee of Faculty of Medicine, Alexandria University
2. Agreement from all participants should be taken in this clinical study by assigning an informed consent
3. Adult end stage renal disease patients maintained on hemodialysis three times a week for at least 3 months with resistant hypertension will be recruited from hemodialysis unit in Alexandria University Hospitals
4. Patients will be screened for resistant hypertension as determined by the mean of mid-week pre-dialysis BP > 140/90 mm Hg, post-dialysis BP > 130/80 mm Hg over a period of one month.
5. A blood sample will be collected for homocysteine measurement at baseline
6. Patients will be randomized using simple randomization technique via computer based program to take one tablet daily containing L-methylfolate and methylcobalamine or no treatment.
7. Patients will be followed over a period of 3 months after which blood pressure measurement and blood sampling would be repeated and compared to baseline values
8. As a measurement of the prognosis of elevated homocysteine, we should follow the development of myocardial infarction, stroke and cardiovascular events for 3 months
9. The appropriate statistical tests will be held according to the study design and parameters to evaluate the significance of the results
10. Results, conclusion, discussion and recommendations will be given

ELIGIBILITY:
Inclusion Criteria:

* Adult end stage renal disease patients maintained on hemodialysis three times a week for at least 3 months with resistant hypertension as determined by pre-dialysis BP > 140/90 mm Hg, post-dialysis BP > 130/80 mm Hg despite the use of three or more drugs

Exclusion Criteria:

* Age > 75 years
* Excessive use of alcohol or smoking
* Severe hepatic impairment
* Acute kidney injury on top of chronic kidney disease
* Pregnant females
* Allergy or intolerance to any component of the formulation
* Medication side effects (methotrexate, theophylline, phenytoin, and cyclosporine) or any drug proven to cause hyperhomocysteinemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
average pre-dialysis blood pressure target of ≤ 140/90 mm Hg or an average post-dialysis blood pressure target of ≤ 130/80 mm Hg | 3 months
  To achieve an average pre-dialysis blood pressure target of ≤ 140/90 mm Hg or an average post-dialysis blood pressure target of ≤ 130/80 mm Hg.
  This should be parallel to lowering of serum homocysteine compared to baseline values

SECONDARY OUTCOMES:
myocardial infarction, stroke and cardiovascular events. | 3 months
  As a measurement of the prognosis patients will be followed up for the development of myocardial infarction, stroke and cardiovascular events for 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan M El-gowelli, PhD, Principal Investigator — Professor of Pharmacology & Toxicology, Alexandria University; Hesham A Elghoneimy, PhD, Principal Investigator — Associate Professor of Internal Medicine, Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Associate Professor of Clinical Pharmacy, Alexandria University; Mohamed S Salem, PharmD, Principal Investigator — Master's student in Clinical Pharmacy and Pharmacy Practice, Alexandria University.
Locations (1):
- Faculty of Pharmacy, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cianciolo G, La Manna G, Coli L, Donati G, D'Addio F, Persici E, Comai G, Wratten M, Dormi A, Mantovani V, Grossi G, Stefoni S. 5-methyltetrahydrofolate administration is associated with prolonged survival and reduced inflammation in ESRD patients. Am J Nephrol. 2008;28(6):941-8. doi: 10.1159/000142363. Epub 2008 Jun 30. PMID 18587236
- [Background] Friedman AN, Bostom AG, Selhub J, Levey AS, Rosenberg IH. The kidney and homocysteine metabolism. J Am Soc Nephrol. 2001 Oct;12(10):2181-2189. doi: 10.1681/ASN.V12102181. PMID 11562419
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Li J, Jiang S, Zhang Y, Tang G, Wang Y, Mao G, Li Z, Xu X, Wang B, Huo Y. H-type hypertension and risk of stroke in chinese adults: A prospective, nested case-control study. J Transl Int Med. 2015 Oct-Dec;3(4):171-178. doi: 10.1515/jtim-2015-0027. Epub 2015 Dec 30. PMID 27847909
- [Derived] Salem MS, Hamdy NA, Elghoneimy HA, El Gowelli HM. Efficacy of L-methylfolate and methylcobalamin in treating resistant hypertension associated with elevated serum homocysteine in hemodialysis patients. BMC Nephrol. 2026 Jan 24. doi: 10.1186/s12882-025-04726-8. Online ahead of print. PMID 41580678